CLINICAL TRIAL: NCT07204834
Title: A Step-Based Physical Activity Intervention in Patients With Heart Failure: The STEP-IN Randomized Controlled Trial
Brief Title: A Physical Activity Program for People With Heart Failure
Acronym: STEP-IN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Department of Physical Education and Sports, Faculty of Sport Sciences, Sport and Health University Research Institute (iMUDS), University of Granada, Spain (Unknown); University Hospital Virgen de las Nieves (Other); Hospital Universitario Clínico San Cecilio (Unknown); Hospital Santa Ana de Motril (Unknown); Mind, Brain and Behaviour Research Centre (CIMCYC) (Unknown); Centro de Investigación Biomédica en Red Fisiopatología de la Obesidad y Nutrición (CIBEROBN), Instituto de Salud Carlos III, Spain (Unknown); Department of Medical BioSciences, Exercise Physiology ResearchGroup, Radboud University Medical Center, Nijmegen, The Netherlands (Unknown); Instituto de Investigación Biosanitaria IBS Granada (Unknown)
Responsible Party: Principal Investigator, Francisco B. Ortega Porcel, Full Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SPID202300X148404IV0
Record Dates: First submitted 2025-09-12; First posted 2025-10-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Exercise; Physical activity; Step; Cadence; Cardiovascular disease; Heart-brain; 6-minute walk test; Walking; Wearable; Fitbit
MeSH Terms: conditions — Heart Failure; Motor Activity; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, participants cannot be blinded to their assigned group. Staff conducting the evaluations will be blinded to the participants' allocation group. Staff conducting statistical analyses for the main outcomes will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): 9-month remotely-monitored, goal-oriented, individualized, step-based physical activity program.
  Interventions: Behavioral: Physical Activity
- Enhanced usual care to manage heart failure (No Intervention): Participants will receive enhanced usual care, consisting of the usual care to manage heart failure (guideline-directed medical therapy) plus an education pamphlet and in-depth evaluations and reports to measure the project outcomes. Specifically, usual care for heart failure generally encompasses optimized treatment titration, patient education and self-management strategies, nurse-led clinical assessments and medication adjustments, monitoring of patient outcomes, and coordinated collaboration with primary care and other specialties.

INTERVENTIONS:
Behavioral: Physical Activity — Participants will be encouraged to progressively increase the number of daily steps (volume) and the number of minutes per day spent at a higher cadence (intensity). To achieve these goals, the investigators will support participants in the intervention group through behavior change techniques. For example, wearable devices and an online platform will be used to monitor the behavior and track progress using simple graphs; participants will be provided with small, individualized goals which will be updated every two weeks based on the activity levels achieved the prior two weeks; standardized WhatsApp messages will be sent to prompt the behavior and face-to-face coaching sessions will be delivered throughout the intervention.
  Participants in this group will also receive enhanced usual care, consisting of the usual care to manage heart failure plus an education pamphlet and in-depth evaluations and reports to measure the project outcomes.
  Other Names: Exercise
  Arms: Physical Activity

SUMMARY:
STEP-IN is a research study that examines the effects of a physical activity program designed to increase the daily steps and cadence of patients with heart failure, compared to standard medical care, on functional capacity and other markers related to heart and brain health.

The primary hypothesis is that participating in the physical activity program for 9 months will improve functional capacity, the primary clinical measure, significantly more than receiving only the standard medical care in people with heart failure. It is also hypothesized that the physical activity program will have positive effects on symptoms and limitations related to heart failure, inflammation, as well as heart and brain health.

DETAILED DESCRIPTION:
Heart failure is associated with disabling symptoms of dyspnea, fatigue, low exercise tolerance, and frequent hospitalizations. Managing heart failure is challenging, as it often coexists with several comorbidities related to cardiovascular- and brain-health (e.g., hypertension, dyslipidemia, cognitive impairment). Physical activity programs represent a promising adjuvant to pharmacological treatments to improve patients' functional capacity, reduce their symptoms, and facilitate long-term physical activity maintenance as patients' exercise tolerance improves. However, few patients with heart failure attend and adhere to traditional structured exercise programs such as cardiac rehabilitation. In response, the overall objective of STEP-IN is to design and test the effectiveness, feasibility and safety of a real-world, individualized step-based physical activity intervention to improve functional capacity, heart failure symptoms and limitations, systemic inflammation and additional heart-brain outcomes in patients with heart failure.

STEP-IN is a two-arm, single-blind multicenter randomized controlled trial. A total of 200 adults with heart failure with reduced (≤40%) or mildly reduced ejection fraction (41-49%) and a II or III NYHA functional class will be enrolled. Participants will be randomized 1:1 to a 9-month step-based physical activity intervention or enhanced usual care. The intervention will leverage wearable devices and a personalized online platform alongside behavior change methods to progressively increase participants' daily step count (volume) and step cadence (intensity), with increments individually planned every 2 weeks. To test the effectiveness of the program all participants will undergo several evaluations at baseline, and 3, 9 and 12 months after randomization, with the main timepoint of interest being from baseline to 9-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure with reduced ejection fraction, HFrEF, i.e., left ventricular ejection fraction ≤40%, or mildly reduced ejection fraction, HFmrEF, i.e., left ventricular ejection fraction 41-49%, confirmed with an echocardiography showing HFrEF or HFmrEF in the last 6 months and having reached stable medication titration (highest tolerated dose) for ≥1 month
* Functional class New York Heart Association (NYHA) II or III, confirmed by the clinical staff
* Age ≥18 years old

Exclusion Criteria:

* Signs or symptoms of decompensated heart failure in the last month
* Uncontrolled arrhythmia
* Limiting angina (grade III or IV)
* Severe symptomatic aortic stenosis
* Persistent symptomatic hypotension
* In the last 3 months: myocardial infarction, revascularization procedure (i.e., percutaneous coronary intervention, coronary artery bypass graft) or insertion of a cardiac device (e.g., implantable cardioverter defibrillator, bi-ventricular pacemaker)
* Comorbid diagnosed conditions that either contraindicate physical activity or may adversely impact adherence to trial procedures, such as active malignancy, major depression or other significant psychiatric disorders, dementia, or significant hearing or visual impairment
* Inability to walk independently (i.e., requires assistive devices for ambulation)
* Already participates in a clinical trial or plans to participate in other interventions that could affect this trial, such as cardiac rehabilitation, during the study period
* Both the participant and caregiver are unable to access a smartphone or internet, or have null technology literacy (i.e., unable to use WhatsApp or a simple Web page)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in functional capacity | Baseline, 3 months, 9 months and 12 months
  The primary outcome is the change in functional capacity measured with a 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Change in patient-perceived heart failure-related symptoms and limitations | Baseline, 3 months, 9 months and 12 months
  Measured with the Kansas City Cardiomyopathy Questionnaire - Clinical Summary Scale (KCCQ-CSS). This is scored on a 0-100 scale, with higher scores indicating better heart failure-related health status (i.e., fewer symptoms and less physical limitation); 0 reflects the worst and 100 the best status.
Change in systemic inflammation | Baseline and 9 months
  Measured with blood-based high-sensitivity C-reactive protein (hs-CRP). Unit: mg/L.
Change in additional pro- and anti-inflammatory markers | Baseline and 9 months
  Additional pro- and anti-inflammatory markers will be measured from a blood sample, e.g., Interleukin-6 (IL-6), Tumor Necrosis Factor-alpha (TNF-α), Interleukin-1 beta (IL-1β), Interleukin-10 (IL-10), and Interleukin-1 Receptor Antagonist (IL-RA), including novel inflammatory biomarkers that may become available up to the time of analysis.
  Unit: pg/mL.
Change in counts of steps | Baseline, 3 months, 9 months (within the last 2 weeks of the intervention) and 12 months
  Measured with a StepWatch accelerometer as the total counts of steps/day.
Change in time spent at light, moderate and vigorous-intensity step cadence | Baseline, 3 months, 9 months (within the last 2 weeks of the intervention) and 12 months
  Measured with a StepWatch accelerometer as minutes/day spent at light, moderate (main interest) and vigorous-intensity step cadence.
Change in peak cadence | Baseline, 3 months, 9 months (within the last 2 weeks of the intervention) and 12 months
  Measured with a StepWatch accelerometer as the minute with the higher number of steps.
Change in 24-hour movement behaviors | Baseline, 3 months, 9 months (within the last 2 weeks of the intervention) and 12 months
  Physical activity (primary behavior of interest), sedentary, and sleep metrics measured with a Matrix Activity Monitor .

OTHER OUTCOMES:
Change in additional heart failure-related patient perceptions | Baseline, 3 months, 9 months and 12 months
  Heart failure-related patient perceptions measured with subscales and individual domains of the Kansas City Cardiomyopathy Questionnaire (KCCQ):
  * Overall Summary Scale (combines symptom, physical limitations, social limitations, and quality of life domains)
  * Self-efficacy Scale. Scores are transformed to a 0-100 scale; higher scores indicate better heart-failure health status.
Change in general cognition | Baseline and 9 months
  Measured with the Montreal Cognitive Assessment (MoCA) total score (1-30).
Change in processing speed | Baseline and 9 months
  Measured by (i) the Trail Making Test Part A (TMT-A), where shorter completion times indicate better performance; and (ii) the Digit Symbol Substitution Test (DSST), with the outcome defined as the total number of correct responses within the time limit (120 sec).
Change in executive function and attentional/Inhibitory control | Baseline and 9 months
  Measured by (i) Trail Making Test Part B (TMT-B), where shorter completion times indicate better performance; (ii) Dimensional Change Card Sort (DCCS), and (iii) the Flanker test, both with computed scores representing accuracy and reaction time.
Change in episodic memory | Baseline and 9 months
  Measured by (i) the free recall item of the Montreal Cognitive Assessment (MoCA), and (ii) the Picture Sequence Memory Test (PSMT), with raw scores indicating memory performance.
Change in brain volume | Baseline and 9 months
  Measured with magnetic resonance imaging using a T1-weighted Magnetization-Prepared Rapid Acquisition Gradient Echo (MPRAGE) structural sequence.
  This outcome will be assessed only in participants without MRI incompatibilities
Change in brain area | Baseline and 9 months
  Measured with magnetic resonance imaging using a T1-weighted Magnetization-Prepared Rapid Acquisition Gradient Echo (MPRAGE) structural sequence.
  This outcome will be assessed only in participants without MRI incompatibilities.
Change in cortical thickness | Baseline and 9 months
  Measured with magnetic resonance imaging using a T1-weighted Magnetization-Prepared Rapid Acquisition Gradient Echo (MPRAGE) structural sequence.
  This outcome will be assessed only in participants without MRI incompatibilities.
Change in brain shapes | Baseline and 9 months
  Measured with magnetic resonance imaging using a T1-weighted Magnetization-Prepared Rapid Acquisition Gradient Echo (MPRAGE) structural sequence.
  This outcome will be assessed only in participants without MRI incompatibilities.
Change in white matter microstructure | Baseline and 9 months
  White matter microstructure will be assessed using diffusion-weighted magnetic resonance imaging, with metrics including mean diffusivity, fractional anisotropy, and tractography-derived measures.
  This outcome will be assessed only in participants without MRI incompatibilities
Change in white matter hyperintensities | Baseline and 9 months
  White matter lesions identified as white matter hyperintensities using 3D T2-weighted Turbo Spin Echo (TSE) Fluid-Attenuated Inversion Recovery (FLAIR) magnetic resonance imaging.
  This outcome will be assessed only in participants without MRI incompatibilities
Change in cerebral blood flow | Baseline and 9 months
  Cerebral blood flow measured with magnetic resonance imaging using the technique of TGSE-pCASL (turbo gradient spin echo-pseudo continuous arterial spin labeling).
  This outcome will be assessed only in participants without MRI incompatibilities
Change in blood-brain barrier permeability | Baseline and 9 months
  Blood Brain Barrier permeability measured by calculating the water exchange rate across the blood-brain barrier using 3D diffusion-prepared arterial spin labelled perfusion magnetic resonance imaging.
  This outcome will be assessed only in participants without MRI incompatibilities
Change in frailty score | Baseline and 9 months
  Frailty score calculated using the Fried Frailty Scale. This scale characterizes frailty as the presence of at least three of the following five components: unintentional weight loss, self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity. Each component in which the participant meets the frailty criterion is scored as 1. Otherwise, it is scored as 0. The scores from the five criteria are summed up to obtain a final score, which is then used to classify the participant according to the following thresholds:
  Frail: ≥3 criteria present. Prefrail: 1-2 criteria. Robust: 0 criteria
Change in anxiety symptoms | Baseline and 9 months
  Reported by participants with the Hospital Anxiety and Depression Scale. The anxiety subscale has 7 items. Each item is rated on a 4-point scale (0-3 points). The total anxiety scores range from 0-21 points. Higher scores mean worse anxiety symptoms.
Change in depression symptoms | Baseline and 9 months
  Reported by participants with the Hospital Anxiety and Depression Scale. The depression subscale has 7 items. Each item is rated on a 4-point scale (0-3 points). The total depression scores range from 0-21 points. Higher scores mean worse depression symptoms.
Change in cardiovascular health score | Baseline and 9 months
  Cardiovascular health score calculated using the total score of Life's Essential 8, and the sub-scores related to health factors and behaviors. The health factors include body mass index, blood lipids, blood glucose and blood pressure. Health behaviors consider physical activity, diet, nicotine exposure and sleep health. It yields a cardiovascular health score based on the unweighted average of all components, ranging from 0 to 100 points. A higher score means better cardiovascular health.
Change in subjective memory decline | Baseline and 9 months
  Reported by participants with the Subjective Memory Decline Scale. It consists of four items assessing self-experienced increasing difficulties in everyday memory, yielding a total score ranging from 0 to 8. Higher scores indicate greater perceived memory decline.
Change in stress | Baseline and 9 months
  Reported by participants with the Perceived Stress Scale (PSS). It consists of 14 items with a five-point response format. A higher score corresponds to a higher level of perceived stress.
Change in loneliness | Baseline and 9 months
  Reported by participants with the UCLA Loneliness Scale. Items are rated using a 4-point Likert-type scale. Total scores range from 10 to 40, with higher scores indicating greater loneliness.
Change in social support | Baseline and 9 months
  Reported by participants with the Multidimensional Scale of Perceived Social Support. The MSPSS is a 12-item self-administered questionnaire that evaluates perceived support from three distinct sources: family, friends, and significant other. Each item is rated on a 7-point Likert scale, with higher scores indicating greater perceived support.
Change in self-esteem | Baseline and 9 months
  Reported by participants with the Rosenberg Self-Esteem Scale. It is a 10-item self-report questionnaire that assesses global self-esteem by capturing individuals' overall sense of self-worth and self-acceptance. Items are rated on a 4-point Likert scale. Total scores range from 10 to 40, with higher scores indicating greater self-esteem.
Change in independence in basic activities of daily living | Baseline and 9 months
  Assessed by a trained health professional, through an interview with the participant, using the Barthel Index. The scale has 10 items covering basic activities of daily living (feeding, bathing, groomig, dressing, continence, toilet use, transfers, mobility and stairs). The total score ranges from 0 to 100 points. Higher scores indicate greater independence in basic activities of daily living.
Change in independence in instrumental activities of daily living | Baseline and 9 months
  Assessed by a trained health professional, through an interview with the participant, using the Lawton and Brody Scale. The scale has 8 items covering instrumental activities of daily living (ability to use the telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for own medication, ability to handle finances). Each item is scored dichotomously (independent = 1, dependent = 0). The total score ranges from 0 to 8 points. Higher scores indicate greater independence in instrumental ADL.
Change in clinical-related measures | Baseline and 9 months
  NYHA category defined by a clinician (I-IV, higher categories denote worse symptoms and limitations), medication prescription
Participants' physical activity enjoyment during the intervention | During the 9-month intervention
  At the end of every month of the intervention, participants will be asked to rate their physical activity enjoyment using a short version of the Physical Activity Enjoyment Scale (PACES). Higher scores indicate greater enjoyment.
  This will be assessed only in participants in the intervention group.
Participants' rating of perceived exertion during the intervention | During the 9-month intervention
  Every two weeks during the intervention, participants will be asked to rate their perceived exertion, thinking about when they were performing step-based physical activities, using the 6-20 Borg scale. Higher scores indicate greater exertion.
  This will be assessed only in participants in the intervention group.
Adherence to and compliance with the intervention | During the 9-month intervention
  Measured based on participants' attendance to the coaching sessions, use of Fitbit and achievement of the goals.
  These will be assessed only in participants in the intervention group
Rate of clinical events during the study | During the study period until the 12-month follow-up
  Based on the incidence of clinical events during the study, i.e., during the 9-month intervention and during the 3-month follow-up (12 months after randomization), including worsening heart failure, hospitalization (cardiovascular and non-cardiovascular related), major adverse cardiovascular events and mortality.
Rate of long-term clinical outcomes | After study completion, an average of 5 and 10 years
  Incidence of clinical events 5 and 10 years after the completion of the study, including hospitalization (cardiovascular and non-cardiovascular related), major adverse cardiovascular events and mortality. This will be measured using structural funds from the research team.
Cost-effectiveness | After study completion, an average of 1 year
  Measured based on analyses of cost-effectiveness. This will be measured using structural funds from the research team.
Social Return on Investment | After study completion, an average of 1 year
  Measured based on analyses of Social Return on Investment (SROI). This will be measured using structural funds from the research team.
Change in natriuretic peptides | Baseline and 9 months
  Measured with peripheral blood-based biomarkers such as N-terminal pro-B-type natriuretic peptide (NT-proBNP).
  Unit: pg/dL.
Change in neurotrophic & growth factors | Baseline and 9 months
  Measured with peripheral blood-based biomarkers such as Brain-Derived Neurotrophic Factor (BDNF).
  Unit: pg/dL.
Change in cholesterol profile | Baseline and 9 months
  Measured with peripheral blood-based biomarkers such as total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides.
  Unit: mg/dL.
Change in glucose profile | Baseline and 9 months
  Measured with peripheral blood-based biomarkers such as Fasting Plasma Glucose. Unit: mg/dL.
Change in glycated hemoglobin | Baseline and 9 months
  Measured with peripheral blood-based glycated hemoglobin (HbA1c). Unit: %.
Change in estimated GFR | Baseline and 9 months
  Estimated as the Glomerular Filtration Rate (eGFR). Unit: mL/min/1.73 m²
Change in markers of renal function | Baseline and 9 months
  Measured with peripheral blood-based creatinine and urea nitrogen (BUN). Unit: mg/dL.
Change in uric acid | Baseline and 9 months
  Measured with peripheral blood-based Uric acid. Unit: mg/dL.
Change in markers of liver function | Baseline and 9 months
  Measured with peripheral blood-based Aspartate aminotransferase, Alanine aminotransferase, Gamma-glutamyl transferase, Alkaline phosphatase, Lactate dehydrogenase, Creatine kinase. Unit: U/L.
Change in total bilirubin | Baseline and 9 months
  Measured with peripheral blood-based Total bilirubin. Unit: mg/dL.
Change in thyrotropin | Baseline and 9 months
  Measured with peripheral blood-based Thyrotropin (TSH). Unit: mIU/L.
Change in parathyroid hormone | Baseline and 9 months
  Measured with peripheral blood-based Parathyroid hormone (PTH, intact). Unit: pg/mL.
Change in markers of coagulation | Baseline and 9 months
  Measured with peripheral blood-based prothrombin time, and activated partial thromboplastin time.
  Unit: seconds
Change in fibrinogen | Baseline and 9 months
  Measured with peripheral blood-based fibrinogen. Unit: mg/dL
Change in electrolytes | Baseline and 9 months
  Measured with peripheral blood-based sodium, potassium, chloride. Unit: mmol/L.
Change in minerals | Baseline and 9 months
  Measured with peripheral blood-based calcium, phosphorus, magnesium. Unit: mg/dL
Change in protein status | Baseline and 9 months
  Measured with peripheral blood-based albumin and total protein. Unit: g/dL
Change in CA 125 | Baseline and 9 months
  Measured with peripheral blood-based Cancer Antigen 125 (CA 125). Unit: U/mL
Change in iron | Baseline and 9 months
  Measured with peripheral blood-based iron. Unit: µg/dL
Change in transferrin | Baseline and 9 months
  Measured with peripheral blood-based transferrin. Unit: mg/dL
Change in transferrin saturation | Baseline and 9 months
  Measured with transferrin saturation index. Unit: %.
Change in Ferritin | Baseline and 9 months
  Measured with peripheral blood-based Ferritin. Unit: ng/mL.
Change in Vitamin D | Baseline and 9 months
  Measured with peripheral blood-based Vitamin D (25 OH). Unit: ng/mL
Change in plasma phosphorylated tau 217 (p-tau217) | Baseline and 9 months
  Measured with blood-based p-tau217. Unit: pg/mL
Change in plasma phosphorylated tau 181 (p-tau181) | Baseline and 9 months
  Measured with blood-based p-tau181. Unit: pg/mL
Change in plasma Aβ42/40 ratio | Baseline and 9 months
  Measured with blood-based amyloid-β 42 to 40 ratio.
Change in plasma neurofilament light (NfL) | Baseline and 9 months
  Measured with blood-based neurofilament light. Unit: pg/mL
Change in additional novel blood-based biomarkers related to heart and brain health | Baseline and 9 months
  The investigators will remain open to assessing novel blood-based biomarkers related to heart and brain health that may become available in the literature up to the time of analysis
Change in handgrip strength | Baseline and 9 months
  Maximal handgrip strength measured at rest using a handheld dynamometer. Higher values indicate better strength.
  Unit: kg.
Change in 30-second chair stand repetitions | Baseline and 9 months
  Number of full stands completed in 30 seconds from a standard chair without using arms. Higher values indicate better lower-body function.
  Unit: repetitions (count).
Change in usual gait speed | Baseline and 9 months
  Usual-pace gait speed measured over a 4.57-meter course from a standing start. Unit: second (m/s).
Change in resting systolic blood pressure | Baseline and 9 months
  Measured with an automated blood pressure monitor (OMRON). Unit: mmHg.
Change in resting diastolic blood pressure | Baseline and 9 months
  Measured with an automated blood pressure monitor (OMRON). Unit: mmHg.
Change in resting heart rate | Baseline and 9 months
  Measured with an automated blood pressure monitor (OMRON). Unit: beats per minute.
Change in body mass index | Baseline and 9 months
  Body mass will be measured using a SECA scale, height will be measured using a SECA height measuring system, body mass index will then be calculated (kg/m2).
Change in waist circumference | Baseline and 9 months
  Measured following standardized procedures with a Lufkin tape measure. Unit: cm.
Changes in biventricular function | Baseline and 9 months
  Measured using resting ultrasound echocardiography with markers such as 2D and 3D ejection fraction, deformation measures, and additional right-ventricular indices.
  Due to logistic constraints, this outcome will only be assessed in participants recruited from the hospitals in Granada city.
Change in cardiac diastolic function | Baseline and 9 months
  Measured using resting ultrasound echocardiography with markers such as E/e' ratio and left atrial strain.
  Due to logistic constraints, this outcome will only be assessed in participants recruited from the hospitals in Granada city.
Change in cardiac dimensions | Baseline and 9 months
  Measured using resting ultrasound echocardiography with markers such as left atrial volume index, and other ventricular and atrial diameters and volumes.
  Unit: mL/m². Due to logistic constraints, this outcome will only be assessed in participants recruited from the hospitals in Granada city.
Change in transcriptomic profile | Baseline and 9 months
  Gene expression analyses will be conducted using RNA blood samples.
Change in epigenomic profile | Baseline and 9 months
  DNA methylation analyses will be conducted using blood samples.
Qualitative usability of the intervention with a custom questionnaire | End of intervention (9 months)
  Measured based on patient perceptions collected using a custom usability questionnaire adapted to the intervention and population, derived from the System Usability Scale. These will be assessed only in participants in the intervention group.
Qualitative usability of the intervention with interviews | End of intervention (9 months)
  Measured based on patient perceptions using semi-structured interviews, such as reported barriers and facilitators.
  These will be assessed only in participants in the intervention group.
Qualitative feasibility of the intervention with interviews | End of intervention (9 months)
  Measured based on patient perceptions using semi-structured interviews, such as ability to engage in the program as intended in daily life.
  These will be assessed only in participants in the intervention group.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Department of Physical Education and Sports, Faculty of Sport Sciences, Sport and Health University Research Institute (iMUDS), University of Granada, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Comarcal Santa Ana de Motril, Motril

IPD SHARING:
Plan to Share IPD: Yes
The protocol and statistical analyses plan will be shared open access.
  Data files including individual participant data (IPD) and their corresponding data dictionaries will be shared under restricted access and upon reasonable request (contact Prof. FB Ortega) due to privacy issues and GDPR regulations.
  IPD will be available for sharing under the "as open as possible, as closed as necessary" principle. The shared data files will be pseudonymized and include only participants who provided informed consent.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD data will be available 12 months after the primary outcome paper is published, upon reasonable request.
Access Criteria: The specific process of data access will be determined at a later stage. Data will be available upon reasonable request to the PI (FB Ortega). The data requests must contain the aim of the research, hypothesis, the specific data being requested, and a data analysis plan. Based on the "as open as possible, as closed as necessary" principle, we will decide whether the data can be shared. A data access committee will be created to discuss and approve any data requests.